CLINICAL TRIAL: NCT01744795
Title: Comparison of CardioQ and Pulmonary Artery Thermodilution Derived Cardiac Output Measurements
Brief Title: CardioQ vs Thermodilution Measurements of Cardiac Output
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasse Moller-Sorensen (Other)
Responsible Party: Sponsor-Investigator, Hasse Moller-Sorensen, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: H-3-2012-063
Record Dates: First submitted 2012-12-04; First posted 2012-12-07 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Comparison of CardioQ and Thermodilution Derived Cardiac Output Measurements
Keywords: cardiac output; thermodilution; esophageal doppler; trending ability
MeSH Terms: interventions — Hemodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- induced changes in hemodynamics (Experimental): Twenty-five patients are planned enrolled. After induction of anesthesia, insertion of the PAC and the CardioQ probe, the patient are placed in the following successive positions: a) supine, b) head-down tilt, c) head-up tilt, d) supine, e) supine with phenylephrine administration f) pace heart rate 80 bpm, g) pace heart rate 110 bpm. CO are measured simultaneously using the CardioQ and thermodilution technique.
  Interventions: Other: induced changes in hemodynamics

INTERVENTIONS:
Other: induced changes in hemodynamics — Twenty-five patients are planned enrolled. After induction of anesthesia, insertion of the PAC and the CardioQ probe, the patient are placed in the following successive positions: a) supine, b) head-down tilt, c) head-up tilt, d) supine, e) supine with phenylephrine administration f) pace heart rate 80 bpm, g) pace heart rate 110 bpm. CO are measured simultaneously using the TEE and thermodilution technique.

SUMMARY:
Minimal invasive monitoring systems of central hemodynamics are gaining increasing popularity. The present study investigates the precision of the esophageal doppler (CardioQ) derived cardiac output and its agreement with pulmonary artery catheter thermodilution (PAC TD) for measuring CO during steady state and with induced hemodynamic changes in patients scheduled for elective cardiac surgery.

DETAILED DESCRIPTION:
Twenty-five patients are planned to be enrolled. After induction of anesthesia, insertion of the PAC and the esophageal-doppler probe, the patient are placed in the following successive positions: a) supine, b) head-down tilt, c) head-up tilt, d) supine, e) supine with phenylephrine administration f) pace heart rate 80 bpm, g) pace heart rate 110 bpm, and CO are measured simultaneously using the CardioQ and PAC TD.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective coronary artery bypass grafting (CABG), who are in stable sinus rhythm, who have a left ventricular ejection fraction > 0.40 measured by transthoracic echocardiography, and who have no significant valve pathology

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Agreement of cardiac output determined with CardioQ, compared with thermodilution | Data are collected in the perioperative period (30min.)
  Data are collected for each patient in the perioperative period. Patients are followed in the first 24 hours. Data will after inclusion of the last data be analysed and appropiate statistics aplied.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rigshospitalet, University of Copenhagen, Copenhagen, Capital Region
  - Department of Cardiothoracic anesthesiology; Rigshospitalet, Copenhagen